CLINICAL TRIAL: NCT04098094
Title: Prevalence of Right Ventricular Dysfunction in Acute Exacerbation of Chronic Respiratory Diseases and Its Impact on Outcomes
Brief Title: Outcomes of RV Dysfunction in Acute Exacerbation of Chronic Respiratory Diseases
Acronym: DVD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Association pour le Développement et l'Organisation de la Recherche en Pneumologie et sur le Sommeil (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A03192-53
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Acute Exacerbation of COPD; Acute Exacerbation of Bronchiectasis; Acute Exacerbation of Asthma; Interstitial Lung Disease; Neuromuscular Diseases; Obesity Hypoventilation Syndrome; Acute Respiratory Failure
MeSH Terms: conditions — Lung Diseases, Interstitial; Neuromuscular Diseases; Obesity Hypoventilation Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational study in patients with chronic respiratory diseases (chronic obstructive pulmonary diseases, bronchiectasis, interstitial lung diseases, neuromuscular diseases, obesity-hypoventilation syndrome...) admitted in intensive care unit for acute respiratory failure. The main objective is to determine the prevalence of right ventricular (RV) dysfunction in this population and to analyze the impact of such a complication on outcomes (survival at day-28, duration of non-invasive or mechanical ventilation, duration of hospital stay). RV function will be assessed by echocardiography at admission, after 3 days and at discharge. Plasma NT-proBNP and troponin levels will be collected.

DETAILED DESCRIPTION:
Observational study in patients with chronic respiratory diseases (chronic obstructive pulmonary diseases, bronchiectasis, interstitial lung diseases, neuromuscular diseases, obesity-hypoventilation syndrome...) admitted in intensive care unit for acute respiratory failure.

Inclusion Criteria:

* Chronic respiratory disease (COPD, ILD, OHS...)
* Admission in ICU for acute respiratory failure
* Patient's non-opposition

Exclusion Criteria:

* Patients < 18 year-old
* Protected patients
* Pregnant women The main objective is to determine the prevalence of right ventricular (RV) dysfunction in this population and to analyze the impact of such a complication on outcomes (survival at day-28, duration of non-invasive or mechanical ventilation, duration of hospital stay). RV function will be assessed by echocardiography at admission, after 3 days and at discharge. Plasma NT-proBNP and troponin levels will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Chronic respiratory disease (COPD, ILD, OHS...)
* Admission in ICU for acute respiratory failure
* Patient's non-opposition

Exclusion Criteria:

* Patients < 18 year-old
* Protected patients
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Observational study in patients with chronic respiratory diseases (chronic obstructive pulmonary diseases, bronchiectasis, interstitial lung diseases, neuromuscular diseases, obesity-hypoventilation syndrome...) admitted in intensive care unit for acute respiratory failure.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-09-19 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Survival | Day 28
  Survival at day 28

SECONDARY OUTCOMES:
Duration of ventilation | Day 28
  Duration of non-invasive ventilation and/or mechanical ventilation

OTHER OUTCOMES:
Duration of hospital stay | Day 28
  Duration of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Demoule, MD, PHD, Principal Investigator — Association pour le Développement et l'Organisation de la Recherche en Pneumologie et sur le Sommeil
Locations (1):
- Service de Pneumologie et Réanimation Médicale, Groupe Hospitalier Pitié Salpêtrière Paris, France, Paris, France

IPD SHARING:
Plan to Share IPD: No